CLINICAL TRIAL: NCT02385318
Title: To Compare Safety and Efficacy of Perrigo's Drug Product Compared to an FDA Approved Drug Product in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-14-019
Record Dates: First submitted 2015-01-30; First posted 2015-03-11 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): Ingenol Mebutate
  Interventions: Drug: Ingenol Mebutate (Perrigo)
- Reference product (Active Comparator): Ingenol Mebutate
  Interventions: Drug: Ingenol Mebutate (Reference)
- Placebo product (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Ingenol Mebutate (Perrigo)
  Other Names: Perrigo product
  Arms: Test Product
Drug: Ingenol Mebutate (Reference)
  Other Names: Reference Listed Drug Product
  Arms: Reference product
Drug: Placebo gel
  Arms: Placebo product

SUMMARY:
The purpose of this study is to compare safety and efficacy of Perrigo's drug product compared to an FDA approved drug product in the treatment of actinic keratosis.

ELIGIBILITY:
Inclusion Criteria

1. Provide written informed consent/assent
2. Healthy male or non-pregnant females, >18 years old
3. Subjects must have clinical diagnosis of actinic keratosis
4. Subjects must be in general good health and free from any clinically significant disease that might interfere with the study evaluations in the opinion of the investigator
5. Subjects must be willing to refrain from using non-approved products on the targeted treatment area during the study period.
6. Subjects should be willing to refrain from using any type of bandage or dressing on the treatment area or apply the gel to open skin wounds, infections, or exfoliative dermatitis.
7. Subjects must be willing and able to comply with the requirements of the study for the duration of the study period.
8. Females of childbearing potential willing to use an acceptable form of birth control

Exclusion

1. Females who are pregnant, nursing, or planning a pregnancy within the study participation period
2. Subjects who are immunocompromised or HIV positive or who have any immune-system disorders including auto-immune disease
3. Subjects who have or had an active herpes infection within 14 days prior to the baseline visit
4. Subjects who have any evidence of carcinoma or any other cancer on the face and scalp
5. Presence of an incompletely healed wound within the treatment area or within 5cm of the treatment area
6. Presence of any skin condition in the treatment area that may be made worse by treatment with the study medication
7. Subjects who have used a tanning salon, tanning booth, sunbathing or have excessive prolonged exposure to the sun 7 days prior to Visit 1/Day 1 (baseline) or planned throughout the study
8. Subjects who plan to use artificial tanners within 5cm of the selected treatment area throughout the study
9. Use of NSAIDs within 7 days from Visit 1/Day 1 (Baseline) or initiation during the trial.
10. Subjects who had select cosmetic or therapeutic procedures within 2cm of the selected treatment area and within 14 days of Visit 1/Day 1 (baseline) or within 10cm of the selected treatment area planned anytime during the study.
11. Subjects who have had or are scheduling elective surgery within 1 month before or after the study period
12. Prior use within 30 days of Visit 1/ Day 1 (baseline) or planned use during the study of immunomodulators, immunosuppressive therapies, interferon, interferon inducers, systemic corticosteroids, and cytotoxic drugs
13. Subjects undergoing treatment or received treatment within 8 weeks of Visit 1/Day 1 (baseline) and within 2cm of the selected area or planned during anytime in the study of: 5-FU, imiquimod, diclofenac, photodynamic therapy used in combination with photosensitizing cream.
14. Subjects who used PUVA or UVB therapy on the face or scalp within 6 months prior to Visit 1/Day 1 (baseline) or are planning to receive PUVA therapy, UVB therapy, or nonprescription UV light sources anywhere on the body during the study.
15. Subjects who have taken systemic chemotherapy medications within the last 6 months prior to Visit 1/Day 1 (baseline) or planned use anytime during the study.
16. Subjects who have undergone resurfacing procedures within the last 6 months prior to Visit 1/Day 1 (baseline) or planned use anytime during the study.
17. Subjects who have been treated within 1 month or planning to receive treatment with systemic retinoids, hyaluronic acid, other medicated actinic keratosis therapy, or topical steroids anywhere on the head during the study.
18. Subject who have a history of hypersensitivity or allergy to any ingredient in the drug product.
19. Use of medicated make-up in the treatment area or significant change in the use of consumer products within 30 days of Visit 1/Day 1 (baseline) and planned use or change throughout the study.
20. Start or change of dose of hormonal treatment within the past 3 months (90 days) or planned start/change throughout the study.
21. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements
22. Participation in any clinical study involving an investigational product, agent, or device in the 30 days prior to Visit 1/Day 1 (baseline) or throughout the study
23. Subjects who have been previously enrolled in this study
24. Employee of the research center or private practice
25. Subjects who in the opinion of the investigator are unlikely to be able to follow the restrictions of the protocol and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: Ingenol Mebutate gel (Perrigo)
- Reference Product: Ingenol Mebutate gel (Reference)
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo Product
Started | 204 | 210 | 105
Completed | 200 | 203 | 99
Not Completed | 4 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Test Product: Ingenol Mebutate
  Ingenol Mebutate (Perrigo)
- Reference Product: Ingenol Mebutate
  Ingenol Mebutate (Reference)
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo Product | Total
Number analyzed (Participants) | 204 | 210 | 105 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.66) | 67.9 (9.91) | 68.4 (9.67) | 67.9 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 54 | 18 | 115
  Male | 161 | 156 | 87 | 404
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 5 | 13
  Not Hispanic or Latino | 198 | 208 | 100 | 506
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 203 | 207 | 104 | 514
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Clearance (Absence) of Actinic Keratosis Lesions as Determined by Visual Inspection of the Investigator
Time Frame: Day 57
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference Product | Placebo Product
Number analyzed (Participants) | 168 | 176 | 83
Participants | 81 | 76 | 10
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — 85% power of success; Yates correction; Equivalence ratio = 1.11, 90% CI 2-sided [-4.38 to 14.44]

ADVERSE EVENTS:
Time Frame: 57 days
Arm/Group | Test Product | Reference Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 1/204 | 0/210 | 0/105
Serious Adverse Events (participants affected / at risk) | 4/204 | 1/210 | 1/105
Other Adverse Events (participants affected / at risk) | 11/204 | 14/210 | 0/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=204) | Reference Product (N=210) | Placebo Product (N=105)
Sudden Death, Probable Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Left Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Worsening of Right Hip Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Gastroenteritis/Food Poisoning (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Sigmoid Diverticulitis/Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=204) | Reference Product (N=210) | Placebo Product (N=105)
APPLICATION SITE PAIN (General disorders) | 11 (11) | 14 (14) | 0 (0)
APPLICATION SITE Pruritus (General disorders) | 7 (7) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02385318/Prot_001.pdf
  • Statistical Analysis Plan (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02385318/SAP_000.pdf